Lipid Biomarkers for Diabetic Heart Disease

PI: Jean Schaffer, MD

Statistical Analysis Plan

Our primary outcome is change (post-intervention - pre-intervention) measures of cardiac function (fractional shortening for systolic function and E' for diastolic function). As a secondary analysis, we will examine the change in C24:0/C16:0 ceramide ratio. Statistical analysis will be performed based on intention to treat. Two-sample t-test or Chi-square test will be used to compare baseline mean values of biomarkers and demographic variables between study groups. ANCOVA will be performed to compare mean change of outcomes between groups adjusting for demographic variables and baseline biomarkers. All statistical tests are two-sided at significance level 0.05.

Updated: 2/1/19